CLINICAL TRIAL: NCT00810368
Title: Carnosine Versus Placebo Treatment Study in Gulf War Illness (GWI)
Brief Title: Treatment Study of Carnosine Versus Placebo in Gulf War Illness (GWI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, James Baraniuk, MD, Professor of Medicine, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-068; USAMRMC PR# W91ZSQ-7149-N602 (Other Grant/Funding Number: CDMRP, DoD); HRPO Log No. A-14542.2 (Other: Human Research Protection Office protocol number)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Persian Gulf Syndrome
Keywords: Carnosine; antioxidant; Persian Gulf War; Gulf War Syndrome; GWI; Gulf War Illness; Exercise; Chronic Fatigue; Fibromyalgia; Veterans; Irritable Bowel Syndrome; Migraine headaches; Neuropathy; Multiple Chemical Sensitivity
MeSH Terms: conditions — Persian Gulf Syndrome; Motor Activity; Fibromyalgia; Irritable Bowel Syndrome; Migraine Disorders; Multiple Chemical Sensitivity | interventions — Carnosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carnosine treatment group (Active Comparator): Carnosine treatment group
  Interventions: Drug: Carnosine
- Placebo control group (Placebo Comparator): Placebo control group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carnosine — 500mg Carnosine x2 daily
  Other Names: Pathway Carnosine supplied by Village Green Apothecary
  Arms: Carnosine treatment group
Drug: Placebo — Microcrystalline cellulose placebo tablets x2 daily
  Other Names: Village Green Apothecary
  Arms: Placebo control group

SUMMARY:
The purpose of this study is to perform a randomized double-blind, placebo-controlled, 12 week study of the effects of carnosine on cognitive, psychometric, autonomic, and muscle strength outcomes in 100 GWI subjects.

DETAILED DESCRIPTION:
Background: Homocarnosine (beta-alanine - gamma-aminobutyric acid) is one of the most abundant dipeptides in the brain. It has important antioxidant properties. Both beta-alanine and GABA are neurotransmitters, suggesting that cleavage of this dipeptide by carnosine dipeptidase 1 (CNDP1) may have important regulatory functions in vivo.

Drug: Homocarnosine is not available. Carnosine (beta-alanine - histidine) is an over-the-counter dietary supplement that shares the antioxidant properties. We proposed that oral carnosine would be absorbed from the gut, cross the blood brain barrier, reduce presumed brain oxidant stress that participated in illness pathology, and improve subject health.

Hypothesis: Carnosine supplementation for 12 weeks by mouth in Gulf War Illness subjects would improve cognitive and other outcomes compared to placebo treatment.

Subjects: Gulf War Illness subjects met 1996 Fukuda criteria for Chronic Multisymptom Illness.

Design: Pilot study. Double blind randomized placebo controlled with comparisons between Week 0 (Baseline, pre-randomization) and Week 12 (end of study) Outcomes: This pilot study included included cognitive testing, magnetic resonance imaging during the 2-back working memory task, self-report of psychometric and other subjective symptoms, tenderness testing by dolormetry, and pain threshold to assess reproducibility in the placebo-treated subjects, and potential treatment effects in the active study drug subjects. The study and each of the outcomes at weeks 0 and 12 are described in detail in the final published paper and in its extensive supplementary on-line materials (Baraniuk JN et al. Glob J Health Sci. 2013 5:69-81. PMID:23618477 PMCID:PMC4209301).

An improvement on accuracy on the 2-back working memory task between 0 and 12 weeks was the primary outcome.

Other evaluations were secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of military enlistment between August 1, 1990 and July 31, 1991, and deployment for 30 consecutive days to:

  * Persian Gulf waters and adjacent land areas,
  * Other global locations, or,
  * U.S. only. 1990-1991 enlistment status:
  * Active duty
  * National Guard
  * Reserves

Exclusion Criteria:

* HIV/AIDS
* Pregnant Women
* Active Duty Military Personnel
* Children
* Incarceration

Ages: 34 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James N Baraniuk, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gray GC, Reed RJ, Kaiser KS, Smith TC, Gastanaga VM. Self-reported symptoms and medical conditions among 11,868 Gulf War-era veterans: the Seabee Health Study. Am J Epidemiol. 2002 Jun 1;155(11):1033-44. doi: 10.1093/aje/155.11.1033. PMID 12034582
- [Background] Baraniuk JN, Casado B, Maibach H, Clauw DJ, Pannell LK, Hess S S. A Chronic Fatigue Syndrome - related proteome in human cerebrospinal fluid. BMC Neurol. 2005 Dec 1;5:22. doi: 10.1186/1471-2377-5-22. PMID 16321154
- [Background] Janssen B, Hohenadel D, Brinkkoetter P, Peters V, Rind N, Fischer C, Rychlik I, Cerna M, Romzova M, de Heer E, Baelde H, Bakker SJ, Zirie M, Rondeau E, Mathieson P, Saleem MA, Meyer J, Koppel H, Sauerhoefer S, Bartram CR, Nawroth P, Hammes HP, Yard BA, Zschocke J, van der Woude FJ. Carnosine as a protective factor in diabetic nephropathy: association with a leucine repeat of the carnosinase gene CNDP1. Diabetes. 2005 Aug;54(8):2320-7. doi: 10.2337/diabetes.54.8.2320. PMID 16046297
- [Background] Chez MG, Buchanan CP, Aimonovitch MC, Becker M, Schaefer K, Black C, Komen J. Double-blind, placebo-controlled study of L-carnosine supplementation in children with autistic spectrum disorders. J Child Neurol. 2002 Nov;17(11):833-7. doi: 10.1177/08830738020170111501. PMID 12585724
- [Result] Baraniuk JN, El-Amin S, Corey R, Rayhan R, Timbol C. Carnosine treatment for gulf war illness: a randomized controlled trial. Glob J Health Sci. 2013 Feb 4;5(3):69-81. doi: 10.5539/gjhs.v5n3p69. PMID 23618477
- See also: Laboratory Website — http://www9.georgetown.edu/faculty/baraniuj/Site/Welcome.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Carnosine Treatment Group: A double blinded placebo controlled study. The pharmacy at Georgetown University Medical Center, will blind the Carnosine. Veterans who meet GWI criteria will be given 500mg Carnosine x2 daily for 12 weeks.
- Placebo Control Group: A double blinded placebo controlled study. The pharmacy at Georgetown University Medical Center, will blind the Placebo. Controls who are aged and gender match and do not meet GWi and other exclusionary criteria microcrystalline cellulose placebo tablets x2 daily for 12 weeks.
Period: Overall Study
Arm/Group | Carnosine Treatment Group | Placebo Control Group
Started | 18 | 15
Completed | 12 | 13
Not Completed | 6 | 2
Not completed — Lost to Follow-up | 4 | 2
Not completed — Lack of Efficacy | 2 | 0

BASELINE CHARACTERISTICS:
Population: Prior 2-back working memory scores in Gulf War Illness were an average of 17 out of 35 correct (5=95%CI). Sample size for a 50% increase in 2-back working memory scores was 13 per group. 10% per month drop out rate was predicted so our aim was to have 36 subjects enter the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Carnosine Treatment Group | Placebo Control Group | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (11.6) | 47.2 (8.7) | 49.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 14 | 10 | 24
Region of Enrollment [Number; unit: participants]
  United States | 18 | 15 | 33

OUTCOME MEASURES:

1. Primary Outcome: Effect of Carnosine Supplementation on Chronic Fatigue Syndrome Severity Scores
Description: CFS Severity Score (Δ ≥ 5 / 36) (Baraniuk et al., 1998; Baraniuk et al., 2000a; Baraniuk, Naranch, Maibach, & Clauw, 2000b). Subjects scored the severity of the 9 CFS criteria (Fatigue, memory/concentration, sore throat, sore lymph nodes, sore muscles, sore joints, headache, sleep disturbances, exertional exhaustion from Fukuda et al. 1994) on a scale of none (score=0), trivial (1), mild (2), moderate (3) and severe (4). The sum was 36.
  Individuals taking carnosine were predicted to show a decrease of ≥ 5 at week 12 compared to week 0, compared to no change for placebo subjects. 2-tailed paired t-tests were used to determine significant incremental changes for individuals in the carnosine group compared to the placebo group.
Time Frame: Weeks 0 and 12
Population: Significant numbers of subjects dropped out of both arms of the study. The primary reason given was perceived lack of efficacy.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Carnosine Treatment Group | Placebo Control Group
Number analyzed (Participants) | 12 | 13
units on a scale | -3.8 [-11.1 to 3.5] | -2.0 [-8.4 to 4.4]
Statistical Analysis 1: Comparison: Carnosine Treatment Group; Description of Power Calculation: The planned sample size completing each arm was based on individual incremental improvements in the primary outcomes of : A) CFS Severity Scores (Baraniuk et al., Annals Allergy Astma Immunol, 1998), B) Instantaneous Fatigue (Kim et al. Journal of Rehab Res Dev, 2010), and C) increased accuracy of 4/35 letters for 2 back working memory task (Owen, Human Brain Mapping, 2005); Test type: Superiority or Other; p = 0.30, t-test, 2 sided — 2-tailed paired Student's t-tests between Week 0 and Week 12 responses (above) were anticipated to show significant benefits with carnosine treatment but no change with placebo. There were no corrections for multiple comparisons in the reported data; Paired t-test
Statistical Analysis 2: Comparison: Placebo Control Group; Test type: Superiority or Other; p = 0.40, t-test, 2 sided

2. Primary Outcome: Subjects With Improved Diarrhea Symptoms
Description: Patients were given questionnaires assessing common symptom complaints of diarrhea.
Time Frame: Weeks 0 and 12
Population: Participants with evaluable data at the end of the study.
Measure: Number; unit: participants
Arm/Group | Carnosine Treatment Group | Placebo Control Group
Number analyzed (Participants) | 7 | 10
participants | 5 | 1
Statistical Analysis 1: Comparison: Carnosine Treatment Group vs Placebo Control Group; Test type: Superiority or Other; p = 0.018, Fisher Exact — Using Fisher's Exact Test, we determined whether there was a significant difference in the number of participants complaining of IBS symptoms; 2 by 2 Fisher's Exact Test

3. Secondary Outcome: Digit Symbol Substitution (WAIS)
Description: Digit Symbol Substitution (WAIS) test (Joy et al., 2000): Subjects were given a table of numerals with matching symbols, and a form with random numerals with open spaces. The objective was to write in as many symbols that corresponded to the random numerals within a 90 second period. Each subject was their own control. The outcome measure was the incremental change in this score between Week 0 and Week 12 (units on a scale). Higher scores indicate better performance.
Time Frame: Difference between Week 0 and Week 12 (end of study)
Population: 2 carnosine subjects had incomplete data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Carnosine Treatment Group | Placebo Control Group
Number analyzed (Participants) | 10 | 13
units on a scale | 10.8 [6.0 to 15.6] | 2.7 [-0.9 to 6.3]
Statistical Analysis 1: Comparison: Carnosine Treatment Group; Test type: Superiority or Other; p = 0.0018, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo Control Group; Test type: Superiority or Other; p = 0.60, t-test, 2 sided

4. Primary Outcome: Incremental Change in Fatigue Score From Baseline to Week 12
Description: Instantaneous Fatigue was scored as none (0) to severe (10) at week 0 and week 12. The difference between the Week 12 minus the Week 0 values was the incremental change. If the incremental change was greater than 0, then the Instantaneous Fatigue was worse at week 12 than week 0. If the incremental change was less than 0, then the Instantaneous Fatigue was improved at week 12 compared to week 0. The total potential range for incremental change was from -10 to +10.
Time Frame: Week 0 and Week 12
Population: Number of participants with evaluable data who completed the study
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Carnosine Treatment Group | Placebo Control Group
Number analyzed (Participants) | 7 | 12
units on a scale | 0.3 [-0.7 to 1.3] | -0.6 [-2.4 to 1.2]

5. Primary Outcome: SF36 Bodily Pain
Description: Incremental change in Medical Outcome Survey Short Form 36 questionnaire (SF36) Bodily Pain score from baseline to week 12. The Medical Outcome Survey Short Form 36 questionnaire (SF36) Bodily Pain score ranges from 0 (very bad bodily pain) to 100 (no bodily pain). The incremental change was the Medical Outcome Survey Short Form 36 questionnaire (SF36) Bodily Pain score at week 12 minus the Medical Outcome Survey Short Form 36 questionnaire (SF36) Bodily Pain score at baseline. The range of scores for incremental change was from -100 to +100. Scores of 0 for Medical Outcome Survey Short Form 36 questionnaire (SF36) Bodily Pain score at baseline and +100 at week 12 indicate an incremental change of 100 - 0 = +100. A score of 100 at baseline for the Medical Outcome Survey Short Form 36 questionnaire (SF36) Bodily Pain score at baseline of +100 at week 12 gives an incremental change of 0 - 100 = -100.
Time Frame: Week 0 and Week 12
Population: Number of participants with evaluable data who completed the study
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Carnosine Treatment Group | Placebo Control Group
Number analyzed (Participants) | 8 | 10
units on a scale | 5.6 [-6.4 to 17.6] | -0.5 [-13.4 to 12.4]
Statistical Analysis 1: Comparison: Carnosine Treatment Group vs Placebo Control Group; Test type: Superiority or Other; p = 0.5, t-test, 2 sided

6. Primary Outcome: Incremental Change in Generalized Anxiety Scale (GAD) Scores From Baseline to Week 12
Description: Each item on the Generalized Anxiety Scale (GAD) scores was scored as none (0), trivial (1), mild (2), moderate (3), or severe (4) and the sum of the 7 items calculated (range 0 to 28). The incremental change between Week 0 and Week 12 was determined for each treatment.
Time Frame: Week 0 and Week 12
Population: Number of participants with evaluable data who completed the study
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Carnosine Treatment Group | Placebo Control Group
Number analyzed (Participants) | 8 | 9
units on a scale | 0.2 [-2.3 to 2.7] | -0.9 [-4.1 to 2.3]
Statistical Analysis 1: Comparison: Carnosine Treatment Group vs Placebo Control Group; Test type: Superiority or Other; p = 0.5, t-test, 2 sided

7. Primary Outcome: Incremental Change in SF36 General Health Between Baseline and Week 12
Description: Incremental change in SF36 General Health score from baseline to week 12. The SF36 General Health score ranges from 0 (very bad General Health) to 100 (very good General Health). The incremental change was the SF36 General Health score at week 12 minus the SF36 General Health score at baseline. The range of scores for incremental change was from -100 to +100. Scores of 0 for SF36 General Health score at baseline and +100 at week 12 indicate an incremental change of 100 - 0 = +100. A score of 100 at baseline for the SF36 General Health score at baseline of +100 at week 12 gives an incremental change of 0 - 100 = -100.
Time Frame: Week 0 and Week 12
Population: Number of participants with evaluable data who completed the study
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Carnosine Treatment Group | Placebo Control Group
Number analyzed (Participants) | 8 | 10
units on a scale | 0.5 [-13.3 to 14.3] | 6.5 [-4.3 to 17.3]
Statistical Analysis 1: Comparison: Carnosine Treatment Group vs Placebo Control Group; Test type: Superiority or Other; p = 0.50, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Carnosine Treatment Group | Placebo Control Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/13
Other Adverse Events (participants affected / at risk) | 2/12 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carnosine Treatment Group (N=12) | Placebo Control Group (N=13)
Elevated CRP Levels (Immune system disorders) | 0 | 1 — At week 6, one subject showed elevated CRP levels (Grade 1, not related). As per protocol, study drug was discontinued for 2 weeks. Hepatitis A, B, and C serologies were negative, and tests normalized. Study drug was restarted with no sequelae.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carnosine Treatment Group (N=12) | Placebo Control Group (N=13)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — A subject with chronic rib pain and tenderness of costochondritis was sent by his primary care physician to a cardiologist. No cardiac pathology was found. This was considered Grade 1, not related.
Hypergammaglobulinemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — One subject had elevated gamma globulins at week 6 (grade 2 adverse event, not related to study drug). The subjects dropped out of the study and was lost to follow-up.

LIMITATIONS AND CAVEATS:
Small sample sizes. No measure of changes in brain carnosine/homocarnosine/GABA.

Subjective outcomes were insensitive to change. Stool consistency needed better scoring system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No